CLINICAL TRIAL: NCT05551468
Title: StayFine: a Personalized Monitoring and Intervention App to Prevent Relapse of Anxiety and Mood Disorders in Youth and Young Adults
Brief Title: StayFine: Personalised Relapse Prevention of Anxiety and Mood Disorders in Youths
Acronym: StayFine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ggz Oost Brabant (Other)
Collaborators: University of Groningen (Other); Amsterdam UMC, location AMC (Other); Accare (Other); RINO ZUID (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 636310007
Record Dates: First submitted 2022-08-29; First posted 2022-09-22 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder; Anxiety Disorders
Keywords: Prevention; Relapse; Child and adolescents psychiatry; Mental Health
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Recurrence; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitoring + Intervention modules (Experimental): Monitoring: Ecological Momentary Assessment (EMA) of affect, thoughts and social company. Optionally with a wearable to measure activity level. Six times per day for two weeks.
  Timepoints: T0-T4.
  Intervention modules: StayFine guided app-based personalised intervention modules. Each individual receives six of eight modules of which three are mandatory and three others are selected based on a personalization procedure.
  Time point: after T0 over the course of three months.
  Interventions: Behavioral: StayFine guided app-based personalised intervention modules; Behavioral: StayFine app-based monitoring
- Monitoring (Active Comparator): Monitoring:Ecological Momentary Assessment (EMA) of affect, thoughts and social company. Optionally with a wearable to measure activity level. Six times per day for two weeks.
  Timepoints: T0-T4.
  Interventions: Behavioral: StayFine app-based monitoring

INTERVENTIONS:
Behavioral: StayFine guided app-based personalised intervention modules — Participants work on guided app-based personalised intervention modules in the StayFine app over the course of three months. The modules are selected by the participant based on shared decision making and a personalized advice. The intervention is based on Preventive Cognitive Therapy (PCT) with elements of Cognitive Behavioral Therapy (CBT) and Positive Psychology. Modules are: psycho education (mandatory), cognitive restructuring (mandatory), positive affect, behavioral activation, exposure, wellness, sleep and a relapse prevention plan (mandatory).
  Arms: Monitoring + Intervention modules
Behavioral: StayFine app-based monitoring — Monitoring six times per day for two weeks in the StayFine app.

SUMMARY:
The current study examines the effectiveness of the StayFine app for relapse prevention of anxiety or depressive disorders in youth using a randomized controlled trial. In addition, ecological momentary assessment (EMA) is used to explore fluctuations in emotions, psychological factors as predictor of the intervention effect and potential differential mechanisms of change. A total of 254 healthy youths remitted from an anxiety and/or depressive disorder, aged 13-21 years old, will be recruited for the study. Participants will be randomized to either 1) use the StayFine app exclusively for monitoring, or 2) use the StayFine app for monitoring and interventions supported by an expert patient. Stratification blocks are of random size and depend on previous episodes (1/2/3 or more) and previous treatment (yes/no). The intervention is based on the well-established Preventive Cognitive Therapy (PCT) for relapse prevention for adults and Cognitive Behavioral therapy adapted for the relapse prevention phase, both supplemented for anxiety and adolescents. In both conditions adolescents monitor their symptoms five times in three years and feedback and treatment advice is given in case of relapse.

The primary outcome will be time to relapse. Secondary outcomes are (core) symptoms of depression and anxiety, number and duration of relapses, global functioning and quality of life. Mediators and moderators will be explored. Exploratory endpoints are monitoring and wearable outcomes.

DETAILED DESCRIPTION:
This study was previously pre-registered in the Netherlands Trial Registry (NTR) on December 15th 2019 with number NL8237. Enrollment started December 16th 2019. This new registry is made because an error was detected in the eligibility criteria listed on the NTR. That registry is taken offline and cannot be updated. Therefore the investigators registered the same study again, but now with updates to correct the wrongly entered information. The previously registered information is available through: https://trialsearch.who.int/Trial2.aspx?TrialID=NL8237

The eligibility criteria and outcomes as defined in the current registry of ClinicalTrials.gov were used from the start of the study and have not been changed during enrollment and recruitment.

In the previous registry the use of a chat-group was mentioned in the intervention. Due to feasibility/planning issues, this was never implemented and therefore this is left out of the current registration. The outcome 'heart rate' is left out as well, because this outcome was not used after a switch in the wearable that measures activity level. Both changes were made before the first participant was enrolled in the study.

The StayFine app runs on the Minddistrict web-based platform that has a CE-certificate. It states that for the Minddistrict platform is in confirmatory with all relevant provisions of Medical Devices Directive 93/42/EEC in conjunction with the following relevant specifications: EN62304:2006+AC:2008; EN-ISO 14971:2012; EN 82304-1:2017.

The StayFine app runs on the Minddistrict web-based platform that has a CE-certificate. It states that for the Minddistrict platform is in conformity with all relevant provisions of Medical Devices Directive 93/42/EEC in conjunction with the following relevant specifications: EN62304:2006+AC:2008; EN-ISO 14971:2012; EN 82304-1:2017.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria at entry of the study:

* Age 13-21 years
* Adolescents who do NOT meet criteria of a current anxiety disorder (separation -, social - or generalized anxiety disorder, specific phobia, panic disorder, agoraphobia) or depressive disorder (major depressive -, persistent depressive -, or disruptive mood dysregulation disorder) based on a semi-structured diagnostic interview (Kiddie Schedule for Affective Disorders and Schizophrenia - lifetime version (K-SADS-PL DSM-5)), but DO meet the criteria for at least one PREVIOUS episode of one or the combination of the above mentioned disorders

Exclusion Criteria:

* A potential subject who currently meets criteria of any of the following mental health problems will be excluded from participation in this study:
* Alcohol or drug misuse
* Previous hypomania and/or mania
* Bipolar disorder
* Previous and/or current psychotic episode

Other exclusion criteria include:

* Only in remission of another anxiety or mood disorder than mentioned above at the inclusion criteria, namely premenstrual dysphoric disorder, depressive disorder due to another medical condition, substance/medication-induced depressive disorder, other specified depressive disorder, unspecified depressive disorder, selective mutism, substance/medication-induced anxiety disorder or anxiety disorder due to another medical condition, other specified anxiety disorder, unspecified anxiety disorder
* only in remission of PTSD or OCD
* ongoing current treatment (more than twice a month) for a mental health disorder including those listed under the inclusion criteria
* no or insufficient mastery of the Dutch language.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 254 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2027-11-21 (Estimated); Study Completion 2027-11-21 (Estimated)

PRIMARY OUTCOMES:
Time to anxiety and/or depressive relapse | up to 36 months (planned: 0, 4, 12, 24, 36 months)
  Time to anxiety and/or depressive relapse over 36 months as assessed by a semi-structured interview: the Kiddie Schedule for Affective Disorders and Schizophrenia - lifetime version (K-SADS-PL DSM-5).

SECONDARY OUTCOMES:
Number of relapses | up to 36 months (planned: 0, 4, 12, 24, 36 months)
  Measured during each semi-structured interview (K-SADS-PL DSM-5). An extra interview may be scheduled if relapse is expected.
Duration of relapse in days | up to 36 months (planned: 0, 4, 12, 24, 36 months)
  Measured during each semi-structured interview (K-SADS-PL DSM-5). An extra interview may be scheduled if relapse is expected.
Global Assessment of Functioning Scale (GAF) | up to 36 months (planned: 0, 4, 12, 24, 36 months)
  Global functioning (0-100). Higher scores mean a better outcome. Measured during each semi-structured interview. An extra interview may be scheduled if relapse is expected.
Revised Children's Anxiety and Depression Scale (RCADS) | up to 36 months (planned: 0, 4, 12, 24, 36 months)
  Anxiety symptoms (0-3 for 31 items). Higher scores mean a worse outcome. Adapted self-report questionnaire RCADS (only including anxiety subscales, total 31 items).
Beck Depression Inventory (BDI) | up to 36 months (planned: 0, 4, 12, 24, 36 months)
  Depressive symptoms (0-3 for 21 items). Higher scores mean a worse outcome.
Dutch version of the EuroQol Questionaire (EQ-5D-Y) | 0, 4, 12, 24, 36 months
  Quality of life (1-3 for 5 items). Higher scores mean a worse outcome. Quality of life (0-100). Higher scores mean a better outcome.

OTHER OUTCOMES:
Descriptives | 0, 4, 12, 24, 36 months
  Age, ethnicity, education level, living situation, previous episodes, previous care, comorbidity, negative life events
Ecological Momentary Assessment (affect, thoughts and social company) | 0, 4, 12, 24, 36 months
  StayFine monitoring outcomes (exploratory endpoint): anxious, sad, angry, stressed, fatigue, experiential avoidance, behavioral avoidance, loneliness, activity costs energy (0-100). Higher scores mean a worse outcome.
  Energetic, relaxed, enthusiastic, happy, pleasurable activity (0-100). Higher scores mean a better outcome. Social company (yes/no).
Wearable data (physical activity) | 0, 4, 12, 24, 36 months
  StayFine monitoring outcomes (exploratory endpoint): the wearable continuously measures acceleration (i.e. movement, vibration and orientation changes in all 3-axes (x,y,z), converted to score estimates of physical activity). The unit of measure is mg (gravitational acceleration). Higher scores mean more activity.
Wearable data (diurnal patterns) | 0, 4, 12, 24, 36 months
  StayFine monitoring outcomes (exploratory endpoint): the wearable continuously measures acceleration (i.e. movement, vibration and orientation changes in all 3-axes (x,y,z), converted to score estimates of physical activity and sleep. This can be converted into diurnal patterns based on time of the day and amount of physical activity and sleep.
Dysfunctional Attitude Scale-17 (DAS-17) | 0, 4, 12, 24, 36 months
  Dysfunctional attitudes (1-7 for 17 items). Higher scores mean a worse outcome.
Positive and negative affect scale (PANAS) | 0, 4, 12, 24, 36 months
  Positive and negative affect (1-5 for 20 items). Higher scores on the 10 positive affect items mean a better outcome. Higher scores on the 10 negative affect items mean a worse outcome.
Behavioral Activation for Depression Scale short form (BADS-SF) | 0, 4, 12, 24, 36 months
  Behavioral Activation (1-7 for 9 items). High scores are consistent with the title of the subscales (e.g., high scores on activation mean more activation and thus a better outcome).
Sleep Reduction Screening Questionnaire (SRSQ) | 0, 4, 12, 24, 36 months
  Sleep (1-3 for 9 items). Higher scores mean a worse outcome.
Perceived Stress Scale (PSS-10) | 0, 4, 12, 24, 36 months
  Stress (0-4 for 10 items). Higher scores mean a worse outcome.
Utrechtse Coping Lijst (UCL) | 0, 4, 12, 24, 36 months
  Coping (1-4 for 47 items). Higher scores mean a better or worse outcome depending on the type of coping (7 in total). For maladaptive strategies higher scores mean a worse outcome, for adaptive strategies higher scores mean a better outcome.
Brief Experiential Avoidance Questionnaire (BEAQ) | 0, 4, 12, 24, 36 months
  Experiential Avoidance (1-6 for 15 items). Higher scores mean a worse outcome.
Dutch Mental Health Continuum-Short Form (MHC-SF) | 0, 4, 12, 24, 36 months
  Flourishing (0-5 for 14 items). Higher scores mean a better outcome.
Adapted Multidimensional Scale of Perceived Social Support (MSPSS-N) | 0, 4, 12, 24, 36 months
  Support (1-7 for 18 items). Higher scores mean a better outcome.
System Usability Scale (SUS) | 0, 4, 12, 24, 36 months
  Usability of StayFine app (1-5 for 10 items). Higher scores mean a better outcome.
Service satisfaction scale (SSS) and 3 questions at the end of an intervention module | 0, 4, 12, 24, 36 months
  Satisfaction with StayFine intervention modules measured using the SSS (1-4 for 4 items). Higher scores mean a better outcome.
  Satisfaction measured using two '0-100' questions at the end of an intervention module. Higher scores mean a better outcome. One open ended question.
(Serious) adverse events | up to 36 months
  If the participants reports an adverse event, it will be registered. During each semi-structured interview, it will be asked as well.
Patient Health Questionnaire for Depression and Anxiety (PHQ4) | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36 months
  A short 4-item screener for core symptoms of anxiety and depression is administered every three months and once extra after the first month (0-3 for 4 items).

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Stikkelbroek, PhD, Principal Investigator — Ggz Oost Brabant
Locations (1):
- GGZ Oost Brabant, Boekel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kooiman BEAM, Robberegt SJ, Albers CJ, Bockting CLH, Stikkelbroek YAJ, Nauta MH. Congruency of multimodal data-driven personalization with shared decision-making for StayFine: individualized app-based relapse prevention for anxiety and depression in young people. Front Psychiatry. 2023 Sep 29;14:1229713. doi: 10.3389/fpsyt.2023.1229713. eCollection 2023. PMID 37840790
- [Background] Robberegt SJ, Brouwer ME, Kooiman BEAM, Stikkelbroek YAJ, Nauta MH, Bockting CLH. Meta-Analysis: Relapse Prevention Strategies for Depression and Anxiety in Remitted Adolescents and Young Adults. J Am Acad Child Adolesc Psychiatry. 2023 Mar;62(3):306-317. doi: 10.1016/j.jaac.2022.04.014. Epub 2022 May 2. PMID 35513189
- [Derived] Robberegt SJ, Kooiman BEAM, Albers CJ, Nauta MH, Bockting C, Stikkelbroek Y. Personalised app-based relapse prevention of depressive and anxiety disorders in remitted adolescents and young adults: a protocol of the StayFine RCT. BMJ Open. 2022 Dec 15;12(12):e058560. doi: 10.1136/bmjopen-2021-058560. PMID 36521888
- See also: Related Info — http://www.stayfine.nl